CLINICAL TRIAL: NCT03481283
Title: A Causative Role for Amylin in Diabetic Peripheral Neuropathy
Status: Recruiting | Type: Observational
Sponsor: Zabeen Mahuwala, MD (Other)
Responsible Party: Sponsor-Investigator, Zabeen Mahuwala, MD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 42732
Record Dates: First submitted 2018-03-01; First posted 2018-03-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Type2 Diabetes; Peripheral Neuropathy
Keywords: Amylin
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Obtaining blood samples and skin biopsy samples to measure amount of amylin present in those tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Three pieces of information lead to the basis for this study:

1. Individuals with Type-2 diabetes commonly develop peripheral neuropathy.
2. Increased production of the hormone amylin occurs in individuals who have Type-2 diabetes.
3. Aggregations of amylin was found in the peripheral vasculature of rats that overexpressed human amylin.

The purpose of this study is to determine whether a correlation exists between the amount of amylin present in the upper extremities of human subjects with Type-2 diabetes and the extent to which symptoms of peripheral neuropathy are expressed in those subjects. The investigators will be testing this by initially collecting blood and skin biopsy samples from subjects, followed by measuring patient sensation and pain responses to heat, cold, and pressure in the upper extremities.

DETAILED DESCRIPTION:
Impaired blood flow through microvessels (arterioles and capillaries) leads to irreversible damage to cells within the affected watershed. In addition to hypertension and age, Type-2 diabetes (DMII) independently contributes to microvascular disease. Distinct from other diabetic complications, the impact of diabetes on neurovascular function has not clearly been shown to correlate with measures of hyperglycemia or peripheral glucose regulation. The pathophysiology underlying the association between type-2 diabetes, vascular injury and neural damage, including CNS parenchymal loss and PNS neuropathy, remains uncertain.

Normally amylin, a byproduct of the synthesis of insulin by pancreatic β-cells, crosses the blood brain barrier and binds to neurons in feeding centers where it is believed to induce anorexic effects. Amylin aggregates are found in microvessels of pancreas, brain, hearts and kidneys of individuals with DMII or obesity. The investigators have demonstrated amylin aggregates in microvessels of peripheral nerves in rats overexpressing human amylin (unpublished). It is unknown whether amylin deposits are a consequence or a trigger of vascular injury, but they are clearly associated and may present a potential target for reducing diabetes-associated microvascular disease. Furthermore, their accumulation in peripheral nerve microvasculature and red blood cells (RBCs) offers possible foci for a peripheral biomarker of diabetes-induced CNS microvascular disease.

Hypothesis: Patients with DMII have significant amylin deposition in the peripheral vasa nervorum and on RBCs that correlates with severity of clinical peripheral polyneuropathy and reduction of peripheral nerve conduction velocities (NCVs); these amylin measures thereby become surrogates of microvascular disease and may serve as metrics of disease severity.

Aim: Obtain serum HbA1c, skin punch biopsy, RBCs, NCVs and clinical sensory examination from forty consenting adults previously diagnosed with DMII. Skin biopsy from volar forearm and red blood cell samples will be processed for amylin deposition.

This pilot study will provide preliminary data to fuel a larger, potentially multi-center, clinical trial investigating the utility of peripheral amylin or RBC amylin as a quantitative biomarker of microvascular disease that would include monitoring the effect of potential therapies. Measuring serum HbA1c will allow for possible correlation to chronic extracellular glucose concentration. Based on our preliminary data from a rat model of type-2 diabetes that expresses human amylin in the pancreas, the investigators anticipate an increased amylin deposition in the skin blood vessels with the progression of type-2 diabetes as measured by sensory examination and NCVs. Although not directly measured in this study, our preliminary data from the analysis of amylin deposition in cerebral blood vessels of patients with type-2 diabetes suggest that APOE 4 carriers, at risk for developing dementia, may have an increased propensity to accumulate amylin deposits in blood vessels. Thus, the ability to easily identify and target a potential driver of microvascular disease may help prevent the devastating effects of the vascular complications of DMII, including cardiovascular disease, retinopathy, nephropathy and dementia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with Type-2 Diabetes.
* Subject shows mild-to-severe peripheral neuropathy, as determined by Nerve Conduction Velocity (NCV) tests.

Exclusion Criteria:

* Subject has not been diagnosed with Type-2 Diabetes.
* Subject shows average, or above average performance on Nerve Conduction Velocity (NCV) tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty patients, age 18 years or older, with previously diagnosed DMII and referred to the Kentucky Neuroscience Institute Neuromuscular Laboratory for nerve conduction velocity studies (NCVs) will be asked to participate in the study. Because this is a pilot study, every effort will be made to select a broad distribution of male and female patients, regardless of ethnicity, who are mildly to severely symptomatic based on NCVs.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Red blood cell amylin level vs severity of peripheral neuropathy | Single time point. Blood sample will be obtained from patient participant immediately after nerve conduction studies are performed.
  RBCs will be harvested from whole blood samples of participants and quantified RBC-bound amylin will be correlated with severity of nerve conduction velocities.
Blood vessel wall amylin deposition vs severity of peripheral neuropathy | Single time point. Skin biopsy will be obtained from patient participant immediately after nerve conduction studies are performed.
  A formalin-fixed 3 mm skin biopsy will be sectioned and stained with an anti-amylin antibody. Level of amylin deposition in blood vessel walls will be correlated with severity of peripheral neuropathy.

SECONDARY OUTCOMES:
Pressure pain threshold vs RBC amylin and blood vessel wall amylin deposition | Participants will undergo pressure test 1 week after providing blood and skin biopsy
  Participants' quantified pain threshold to applied pressure over the thenar eminence using a pressure algometer will be correlated to both RBC amylin and blood vessel wall amylin deposition.
Cold pressor test vs RBC amylin and blood vessel wall amylin deposition | Participants will undergo cold pressor test 1 week after providing blood and skin biopsy
  Participants' quantified pain threshold to a cold water bath (1 deg C) emmersion of their non-dominant forearm will be correlated to both RBC amylin and blood vessel wall amylin deposition.
Heat thermode test vs RBC amylin and blood vessel wall amylin deposition | Participants will undergo heat thermode test 1 week after providing blood and skin biopsy
  Participants' quantified pain threshold to a thermode placed on the dominant forearm will be correlated to both RBC amylin and blood vessel wall amylin deposition.

CONTACTS AND LOCATIONS:
Overall Officials: John T Slevin, M.D., M.B.A., Principal Investigator — University of Kentucky Department of Neurology; Zabeen Mahuwala, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - UK Robert Straus Behavioral Science Laboratory, Lexington, Kentucky
  - University of Kentucky - Kentucky Neuroscience Institute, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT03481283/Prot_000.pdf